CLINICAL TRIAL: NCT06096337
Title: A Prospective Randomized Multicenter Global Study Comparing Pulsed Field Ablation (PFA) Versus Anti-Arrhythmic Drug (AAD) Therapy as a First Line Treatment for Persistent Atrial Fibrillation
Brief Title: Pulsed Field Ablation (PFA) vs Anti-Arrhythmic Drug (AAD) Therapy as a First Line Treatment for Persistent Atrial Fibrillation
Acronym: AVANT GUARD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF303
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Insertable Cardiac Monitor; Pulsed Field Ablation; Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases | interventions — Drug Delivery Systems; Sotalol; Propafenone; dofetilide; Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulsed Field Ablation (PFA) (Experimental): Pulsed Field Ablation (PFA) is used as the initial treatment for subjects with persistent atrial fibrillation (AF)
  Interventions: Device: FARAPULSE™ Pulsed Field Ablation (PFA) System
- Anti-Arrhythmic Drug (AAD) (Active Comparator): Anti-Arrhythmic Drug (AAD) is used as the initial treatment for subjects with persistent atrial fibrillation (AF)
  Interventions: Drug: Anti-Arrhythmic Drug (AAD): Flecainide, Sotalol, Propafenone, Dofetilide, and Dronedarone

INTERVENTIONS:
Device: FARAPULSE™ Pulsed Field Ablation (PFA) System — Subjects will undergo a pulsed field ablation procedure using the FARAPULSE™ Pulsed Field Ablation (PFA) System for the isolation of pulmonary veins and posterior wall.
  Arms: Pulsed Field Ablation (PFA)
Drug: Anti-Arrhythmic Drug (AAD): Flecainide, Sotalol, Propafenone, Dofetilide, and Dronedarone — Anti-Arrhythmic Drugs (AADs) including, Flecainide, Sotalol, Propafenone, Dofetilide, and Dronedarone will be prescribed and monitored in accordance with local clinical practice and already established guideline-directed therapy for patients with persistent atrial fibrillation (AF).
  Arms: Anti-Arrhythmic Drug (AAD)

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of pulsed field ablation as a first-line ablation treatment for subjects with persistent atrial fibrillation as compared to subjects who received an initial treatment with anti-arrhythmic drugs.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center, global, pivotal Investigational device exemption (IDE) study. Subjects with persistent atrial fibrillation will be randomized or assigned to either pulsed field ablation (PFA) or Versus Anti-Arrhythmic Drug (AAD) treatment.

Once randomization is complete, additional subjects will be enrolled and sequentially assigned to receive PFA treatment to fulfill the number of subjects required for the Primary Safety Endpoint assessment. These additional subjects are referred to as PFA Assigned (Non-Roll-In) Subjects.

Subjects randomized or assigned to PFA treatment will undergo percutaneous ablative pulmonary vein isolation (PVI) and left atrial posterior wall isolation (PWI) using the FARAWAVE™ PFA Catheter (first-line ablation cohort).

Subjects randomized to AAD treatment will be prescribed and monitored in accordance with local clinical practice and already established guideline-directed therapy for patients with persistent atrial fibrillation (AF). In the case of clinical inefficacy, the AAD dose will be up-titrated to the maximum tolerated dose. Thereafter, a change to a second or to a third AAD should be undertaken, insofar as the subject remains within the blanking period, with the goal to completely suppress AF episodes ≥ 30 seconds in duration. If AAD treatment is proven to be ineffective or intolerable outside of the blanking period, subjects can undergo subsequent ablation therapy and be considered part of the "delayed ablation cohort".

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age, or older if specified by local law
2. Have symptomatic persistent AF, confirmed by both:

   a. Documentation, within 180 days of randomization, or treatment assignment for roll-in subjects, of either: i. A 24-hour continuous ECG recording (from any regulatory cleared rhythm monitoring device) confirming continuous AF, OR ii. Two ECGs (from any regulatory cleared rhythm monitoring device) showing continuous AF taken at least 7 days apart b. Documentation, such as physician note, of persistent continuous AF for > 7 days and ≤ 365 days
3. Willing and capable of providing informed consent
4. Willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center
5. Willing to receive LUX-Dx™ insertable cardiac monitor (ICM) during the study or already has a LUX-Dx™ ICM that was inserted ≤ 6 months(i.e., within 180 days of consent

Exclusion Criteria:

1. Treated with AAD (Class I or III) ≤ 6 months (i.e., within 180 days) before enrollment,

   1. More than 7-day history of therapeutic AAD use (Class I or III), or
   2. ≥ 24 hours amiodarone, i Note Pill-in-the-pocket AAD use, is permitted.
2. Treated with AAD ( Class I or III) > 6 months (i.e., more than 180 days) before enrollment and experienced AAD failure (adverse drug effects or frequent AF episodes)
3. Contraindication to, or unwillingness to use, AADs (Class I and III, excluding amiodarone)
4. Contraindication to PFA treatment
5. Contraindication to, or unwillingness to use, systemic anticoagulation, or acceptable alternatives, pre-, intra-, and post-procedure to achieve adequate anticoagulation.
6. Any of the following atrial conditions:

   1. Left atrial (LA) anteroposterior diameter ≥ 5.5 cm, or, if LA diameter not available, non-indexed volume >100 ml, as documented by physician note or imaging (Note: if both values are available, only the LA diameter will be used to confirm eligibility criteria)
   2. Any prior atrial endocardial, epicardial or surgical ablation procedure for arrhythmia, other than right sided cavotricuspid isthmus ablation or for right sided supraventricular tachycardia
   3. Current atrial myxoma
   4. Any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
   5. Current left atrial thrombus
7. Any of the following cardiovascular conditions:

   1. History of sustained ventricular tachycardia or any ventricular fibrillation
   2. AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
   3. Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, interatrial baffle, atrial septal patch, atrial septal defect closure device, or patent foramen ovale occluder
   4. Valvular disease that is any of the following: i. Symptomatic, ii. Causing or exacerbating congestive heart failure, iii. Associated with abnormal left ventricular (LV) function or hemodynamic measurements
   5. Hypertrophic cardiomyopathy
   6. Cardiac amyloidosis
   7. Any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty
   8. Any inferior vena cava (IVC) filter, known inability to obtain vascular access or other contraindication to femoral access
   9. Rheumatic heart disease
   10. Congenital heart disease with any clinically significant residual anatomic or conduction abnormality
   11. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
8. Any of the following conditions identified during screening assessments

   1. Heart failure associated with New York Heart Association (NYHA) Class IV
   2. Left Ventricle Ejection Fraction (LVEF) < 40%
   3. Uncontrolled hypertension (Systolic Blood Pressure > 160 mmHg or Diastolic Blood Pressure > 95 mmHg on two (2) BP measurements during screening
9. Any of the following events 90 days prior to randomization (or Index procedure for PFA Assigned or roll-in subjects):

   1. Myocardial infarction (MI), unstable angina or coronary intervention
   2. Cardiac surgery
   3. Heart failure hospitalization
   4. Pericarditis or symptomatic pericardial effusion
   5. Gastrointestinal bleeding
   6. Stroke, TIA, or intracranial bleeding
   7. Non-neurologic thromboembolic event
   8. Carotid stenting or endarterectomy
10. Known coagulopathy disorder (e.g., von Willbrand's disease, hemophilia)
11. Unwillingness to receive, or unable to tolerate, a subcutaneous, chronically inserted LUX-Dx™ ICM device
12. Women of childbearing potential who are pregnant, lactating, not using a reliable form of contraception, or who are planning to become pregnant during the anticipated study period
13. Body Mass Index (BMI) > 45
14. Solid organ or hematologic transplant, or currently being evaluated for a transplant
15. Any prior history or current evidence of hemi-diaphragmatic paralysis or paresis
16. Severe lung disease, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
17. Severe pulmonary hypertension during screening assessment
18. Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
19. Active malignancy at enrollment (other than cutaneous basal cell or squamous cell carcinoma)
20. Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
21. Known active systemic infection
22. Uncontrolled diabetes mellitus or a recorded HgbA1c > 8.0% in the 90 days prior to randomization (or Index procedure for PFA Assigned or roll-in subjects)
23. Untreated diagnosed obstructive sleep apnea with apnea hypopnea index classification of severe (>30 pauses per hour)
24. Predicted life expectancy less than one (1) year
25. Currently enrolled in another investigational study or registry that would directly interfere with this study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility
26. Health conditions that, in the investigator's medical opinion, would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation
27. Has operational LUX-Dx ICM that was inserted more than 6 months (i.e., >180 days) prior to enrollment
28. Has operational ICM other than a LUX-Dx ICM and does not express a willingness to receive a LUX-Dx ICM for the study
29. Individuals who may require an ablation, besides the PV and PW, in the left atrium including, but not limited to, those with Left-Sided Atrioventricular Reentrant Tachycardia (AVRT), Left-Sided Atrial Tachycardia (AT), or Atypical Left-Sided Atrial Flutter.
30. AAD (Class I and III) Drug Naïve Subjects (as defined in criterion #1 and #2), who are PFA Assigned (Non-Roll-in), PFA randomized, or Roll-in with a CHA2DS2-VASc Score ≥ 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2028-02-03 (Estimated)

PRIMARY OUTCOMES:
Rate of randomized PFA or PFA Assigned subjects with PFA System inserted into the body, during the index or repeat PFA procedure during blanking period, with device or procedure-related Composite Adverse Events that is serious. | 12-Months
  Defined Composite Adverse Events:
  Day 0 through Day 7:
  * Gastric motility / pyloric spasm disorders
  * Heart block
  * Myocardial infarction
  * Peripheral or organ thromboembolism
  * Pulmonary edema
  * Stroke/ Cerebrovascular accident (CVA)
  * Transient ischemic attack (TIA)
  * Unresolved phrenic nerve palsy / paresis
  * Vascular access complications
  Day 0 through Day 30:
  * Cardiac tamponade / perforation
  * Cardiovascular or pulmonary adverse event
  * Death
  * Pericarditis
  Day 0 through Month 12:
  * Atrio-esophageal fistula
  * Pulmonary vein stenosis
Rate of intent to treat subjects with treatment success from the pulse field ablation treatment and Anti-Arrhythmic Drug treatment. | 12-Months
  Defined Treatment Success:
  PFA and AAD Treatment Arms:
  • Amiodarone freedom from randomization to Month 12 unless previously an acute or chronic primary effectiveness failure.
  PFA Treatment Arm:
  • Acute Success - Isolation of attempted pulmonary veins and left atrial posterior wall during blanking period with PFA system
  And
  Chronic Success: Freedom during blanking period to Month 12 of:
  * Occurrence ≥ 1 hr of asymptomatic or ≥ 30 sec of symptomatic Atrial Fibrillation (AF), Atrial Flutter (AFL), or Atrial Tachycardia (AT)
  * Any re-ablation for AF, AFL, or AT
  * Any electrical cardioversion for AF, AFL, or AT
  * Any Class I or III AAD use
  AAD Treatment Arm:
  Acute Success - Ablation not performed in blanking period
  Chronic Success - Freedom after blanking period through Month 12 of:
  * Detectable occurrence ≥ 1 hr of asymptomatic or ≥ 30 sec of symptomatic AF, AFL, or AT
  * Electrical cardioversion for AF, AFL, or AT
  * Any ablation for AF, AFL, or AT

SECONDARY OUTCOMES:
Atrial fibrillation burden between the pulsed field ablation and anti-arrhythmic drug arm, as the LUX-Dx Insertable Cardiac Monitor measures and defined as proportion of time individual spends in AF during a period (expressed as a percentage). | 12, 24, and 36 Months
  Atrial Fibrillation (AF) burden, measured by the LUX-Dx Insertable Cardiac Monitor (ICM) between the 2 randomized groups:
  * Pulsed Field Ablation (PFA) as initial treatment for subjects with persistent AF
  * Anti-Arrhythmic Drug (AAD) as initial treatment for subjects with persistent AF
  Defined AF Burden is proportion of AF time during a period (expressed as a percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Wazni, M.D., Principal Investigator — The Cleveland Clinic
Locations (62):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Scripps Memorial Hosptial, La Jolla, California
  - Stanford University Medical Center, Palo Alto, California
  - Cardiology Associates Medical Group, Inc, Ventura, California
  - HCA Florida Mercy Hospital, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - St. John's Hospital, Springfield, Illinois
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - Mercy Hospital Medical Center-Hospital, West Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Southcoast Physicians Group, Fall River, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic Foundation-Hospital, Rochester, Minnesota
  - Catholic Medical Center, Manchester, New Hampshire
  - Valley Hospital, Paramus, New Jersey
  - Northwell Health, Bay Shore, New York
  - Kaleida Health, Buffalo, New York
  - Weill Cornell Medical University, New York, New York
  - Good Samaritan - Suffern, Suffern, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - York Hospital, York, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Orion Medical, Houston, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - Chippenham & Johnston-Willis Hospital (CJW), Richmond, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (3):
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital-Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
- Medizinische Univ.-Kliniken Graz-Hospital, Graz, Austria
- St. Jan, Bruges, Belgium
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
- Klinicki Bolnicki Centar Split, Split, Croatia
- CHU Grenoble - Hopital Michallon, Grenoble, France
- Germany (2):
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Italy (4):
  - AOU delle Marche - PO GM Lancisi, Ancona, AN
  - Centro Cardiologico Monzino, Milan, MI
  - Maria Cecilia Hospital SPA, Cotignola, RA
  - Fondazione PTV - Policlinico Tor Vergata, Roma
- National Heart Centre Singapore, Singapore, Singapore
- Hospital Universitario La Fe, Valencia, Spain
- Taipei Veterans General Hospital-Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No